CLINICAL TRIAL: NCT02602080
Title: Patient Recovery After Orthopedic Surgery Under Nerve Blocks With Sedation in Foot and Ankle Patients (FA) and Nerve Block With Either Sedation or General Anesthesia (GA) in Total Shoulder Arthroplasty (TSA) Patients. A Pilot Study
Brief Title: Post- Surgery Recovery: Nerve Blocks w/ Sedation vs. Nerve Block w/ Either Sedation/Gen. Anesthesia
Status: Completed | Type: Observational
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-397
Record Dates: First submitted 2015-11-04; First posted 2015-11-11 (Estimated); Results first posted 2019-02-04 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Nausea; Emesis
MeSH Terms: conditions — Nausea; Vomiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- FA patients under popliteal block + spinal + sedation: Foot and ankle patients under popliteal block+ spinal+ sedation
- TSA patients under brachial plexus block + general (LMA): Total shoulder arthroscopy patients under brachial plexus block + general (LMA)
- TSA patients under brachial plexus block + sedation: Total shoulder arthroplasty patients under brachial plexus block + sedation

SUMMARY:
Nausea after surgery may negatively influence patient satisfaction, may delay discharge, and cause unexpected hospital admissions. The trend toward ambulatory surgery has increased the focus on postoperative nausea, but published evidence is not based on standardized criteria for assessment. Therefore, the results for postoperative nausea are very diverse, especially reports on nausea incidence after regional anesthesia, i.e. spinal anesthesia. When peripheral nerve blocks have been applied for postoperative pain control, they significantly reduce postoperative pain, opioid consumption and side effects; patients receiving general anesthesia (GA) and nerve blocks are thought likely to have less nausea than patients receiving GA alone. This study is a pilot study looking at the incidence and intensity of nausea after orthopedic surgery under nerve blocks in foot and ankle (FA) patients and under nerve blocks with either sedation or GA in total shoulder arthroplasty (TSA) patients. The results of this study will help power a future randomized controlled trial, comparing the incidence and intensity of nausea in FA patients receiving GA through laryngeal mask airway (LMA) versus spinal anesthesia.

DETAILED DESCRIPTION:
Nausea after surgery may negatively influence patient satisfaction, may delay discharge, and cause unexpected hospital admissions. The trend toward ambulatory surgery has increased the focus on postoperative nausea, but published evidence is not based on standardized criteria for assessment. Therefore, the results for postoperative nausea are very diverse, especially reports on nausea incidence after regional anesthesia, i.e. spinal anesthesia. This is due to varying data sources, such as nurse notes and/or patient reports, and a lack of a consistent antiemetic and pain medication protocol. The results of this study will help power a future randomized controlled trial, comparing the incidence and intensity of nausea in FA patients receiving GA through laryngeal mask airway (LMA) versus spinal anesthesia.

When peripheral nerve blocks have been applied for postoperative pain control, they significantly reduce postoperative pain, opioid consumption and side effects; patients receiving GA and nerve blocks are thought likely to have less nausea than patients receiving GA alone, due a reduction in pain leading to reduction in need for emetogenic opioids.

This study is a pilot study looking at the incidence and intensity of nausea after orthopedic surgery under nerve blocks in foot and ankle (FA) patients and under nerve blocks with either sedation or GA in total shoulder arthroplasty (TSA) patients. At the author's institution, TSA is commonly performed with a brachial plexus block and either GA or intravenous sedation. TSA patients represent a model system for the effect of GA on nausea among patients receiving nerve blocks.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery
* Age 18-99
* Patients who are capable to provide informed consent and answer questions in English,
* For FA patients: Planned neuraxial anesthesia + nerve block for postsurgical analgesia,
* For TSA patients: Planned brachial plexus nerve block + either general anesthesia or IV sedation.

Exclusion Criteria:

* Incapable to provide informed consent
* Contraindications for regional or LMA anesthesia (anticoagulation, infection at injection site)
* Anticipated difficult airway
* Body mass index>35
* Anticipated surgical procedure time less than 1 hour or more than 4 hours,
* History of severe postoperative nausea and/or vomiting
* American Society of Anesthesiologists physical status classification >3
* Neuropathy
* Pregnant or nursing women
* Chronic opioid use (daily use of opioids one month prior to surgery/ patients requiring chronic pain interventions)
* Prone position planned for surgery
* Obstructive sleep apnea
* Known allergy/sensitivity to any study medications

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective orthopedic surgery for foot and ankle or total shoulder replacement that are within the age limit and meet eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2015-12; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Ya Deau, MD, PhD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 55 patients were enrolled in the study based on the anesthesia they will be receiving and their surgical type. Patients weren't excluded prior to group assignment. Patients were excluded if protocol deviations occurred, pending the severity of the deviation.
Period: Overall Study
Arm/Group | FA Patients Under Popliteal Block + Spinal + Sedation | TSA Patients Under Brachial Plexus Block + General (LMA) | TSA Patients Under Brachial Plexus Block + Sedation
Started | 21 | 16 | 18
Completed | 15 | 15 | 15
Not Completed | 6 | 1 | 3
Not completed — Protocol Violation | 6 | 1 | 3

BASELINE CHARACTERISTICS:
Population: Patients contributed baseline units by patient report (history of PONV, motion sickness, smoking status) and by granting access to their charts (age, gender, race, ethnicity, ASA status, BMI).
Groups:
- Total: Total of all reporting groups
Arm/Group | FA Patients Under Popliteal Block + Spinal + Sedation | TSA Patients Under Brachial Plexus Block + General (LMA) | TSA Patients Under Brachial Plexus Block + Sedation | Total
Number analyzed (Participants) | 15 | 15 | 15 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 3 | 5 | 20
  >=65 years | 3 | 12 | 10 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (15) | 71 (8) | 68 (9) | 65 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 8 | 31
  Male | 3 | 4 | 7 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 13 | 14 | 14 | 41
  Unknown or Not Reported | 1 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0
  White | 10 | 14 | 13 | 37
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 15 | 45
BMI [Mean (Standard Deviation); unit: kg/m^2] | 25 (4) | 26 (4) | 29 (3) | 27 (4)
American Society of Anesthesiologists (ASA) physical status (PS) [Count of Participants; unit: Participants]
  ASA PS I (normal healthy patient) | 4 | 1 | 2 | 7
  ASA PS II (patient with mild systemic disease) | 11 | 13 | 10 | 34
  ASA PS III (patient with severe systemic disease) | 0 | 1 | 3 | 4
Current smoking status [Count of Participants; unit: Participants]
  Yes (smoker) | 2 | 1 | 1 | 4
  No (non-smoker) | 13 | 14 | 14 | 41
History of post-operative nausea and vomiting (PONV) [Count of Participants; unit: Participants]
  Yes | 3 | 2 | 4 | 9
  No | 12 | 12 | 10 | 34
  No prior surgery | 0 | 1 | 1 | 2
Anesthesia Time [Mean (Standard Deviation); unit: min] | 169 (51) | 132 (11) | 133 (18) | 145 (27)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Nausea 1 Hour After Post-anesthesia Care Unit (PACU) Admission
Description: Yes/no response to whether patient had nausea in the PACU 1 hour after admission. If yes, investigators will seek out intensity
Time Frame: 1 hour after surgery
Population: Patients receiving either block+spinal+sedation for foot and ankle surgery or block+general or block+sedation for total shoulder arthroscopy
Measure: Count of Participants; unit: Participants
Arm/Group | FA Patients Under Popliteal Block + Spinal + Sedation | TSA Patients Under Brachial Plexus Block + General (LMA) | TSA Patients Under Brachial Plexus Block + Sedation
Number analyzed (Participants) | 15 | 15 | 15
Participants
  Yes | 1 | 0 | 1
  No | 14 | 15 | 14

2. Primary Outcome: Number of Participants With Nausea
Description: Yes/no question. If yes, the investigators will then seek intensity of nausea.
Time Frame: Average 2 hours after surgery (at discharge from the recovery room after surgery)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | FA Patients Under Popliteal Block + Spinal + Sedation | TSA Patients Under Brachial Plexus Block + General (LMA) | TSA Patients Under Brachial Plexus Block + Sedation
Number analyzed (Participants) | 15 | 15 | 15
Participants
  Yes | 2 | 0 | 2
  No | 13 | 15 | 13

3. Primary Outcome: Intensity of Nausea
Description: On an 11 grade Likert scale (0=no nausea, 10=worst possible nausea)
Time Frame: 1 hour after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | FA Patients Under Popliteal Block + Spinal + Sedation | TSA Patients Under Brachial Plexus Block + General (LMA) | TSA Patients Under Brachial Plexus Block + Sedation
Number analyzed (Participants) | 15 | 15 | 15
Participants
  0 | 14 | 15 | 14
  1 | 0 | 0 | 0
  2 | 0 | 0 | 1
  3-7 | 0 | 0 | 0
  8 | 1 | 0 | 0
  9-10 | 0 | 0 | 0

4. Primary Outcome: Intensity of Nausea
Description: On a 11 grade Likert scale (0=no nausea, 10=worst possible nausea)
Time Frame: 2 hours after surgery
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | FA Patients Under Popliteal Block + Spinal + Sedation | TSA Patients Under Brachial Plexus Block + General (LMA) | TSA Patients Under Brachial Plexus Block + Sedation
Number analyzed (Participants) | 15 | 15 | 15
Participants
  0 | 13 | 15 | 13
  1 | 0 | 0 | 1
  2-4 | 0 | 0 | 0
  5 | 1 | 0 | 1
  6-8 | 0 | 0 | 0
  9 | 1 | 0 | 0
  10 | 0 | 0 | 0

5. Secondary Outcome: Antiemetic Consumption
Description: Yes/no question if antiemetic consumption occured.
Time Frame: Duration of stay in recovery room after surgery (average 2 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | FA Patients Under Popliteal Block + Spinal + Sedation | TSA Patients Under Brachial Plexus Block + General (LMA) | TSA Patients Under Brachial Plexus Block + Sedation
Number analyzed (Participants) | 15 | 15 | 15
Participants
  Yes | 2 | 0 | 0
  No | 13 | 15 | 15

6. Secondary Outcome: Number of Participants With Emesis
Description: Yes/no question. If yes, the investigators will then seek intensity of emesis
Time Frame: 1 hour after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | FA Patients Under Popliteal Block + Spinal + Sedation | TSA Patients Under Brachial Plexus Block + General (LMA) | TSA Patients Under Brachial Plexus Block + Sedation
Number analyzed (Participants) | 15 | 15 | 15
Participants
  Yes | 0 | 0 | 0
  No | 15 | 15 | 15

7. Secondary Outcome: Number of Participants With Emesis
Description: Yes/no question. If yes, the investigators will then seek intensity of emesis
Time Frame: Average 2 hours after surgery (at discharge from the recovery room after surgery)
Measure: Count of Participants; unit: Participants
Arm/Group | FA Patients Under Popliteal Block + Spinal + Sedation | TSA Patients Under Brachial Plexus Block + General (LMA) | TSA Patients Under Brachial Plexus Block + Sedation
Number analyzed (Participants) | 15 | 15 | 15
Participants
  Yes | 0 | 0 | 0
  No | 15 | 15 | 15

8. Secondary Outcome: Number of Participants Satisfied With Anesthesia
Description: Lowest satisfaction score on a 11 grade Likert scale (0=no satisfaction, 10=maximal satisfaction).
Time Frame: PACU before discharge, an average of 2 hours
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | FA Patients Under Popliteal Block + Spinal + Sedation | TSA Patients Under Brachial Plexus Block + General (LMA) | TSA Patients Under Brachial Plexus Block + Sedation
Number analyzed (Participants) | 15 | 15 | 15
score on a scale | 10 [10 to 10] | 10 [10 to 10] | 10 [9 to 10]

9. Secondary Outcome: Patients Receiving Opioids in the PACU
Description: Yes/no for patients that were given opioids for pain management in the PACU. If opioids were consumed, the oral morphine equivalents for the patients taking opioids was totaled.
Time Frame: PACU stay before discharge (average 2 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | FA Patients Under Popliteal Block + Spinal + Sedation | TSA Patients Under Brachial Plexus Block + General (LMA) | TSA Patients Under Brachial Plexus Block + Sedation
Number analyzed (Participants) | 15 | 15 | 15
Participants
  Yes | 4 | 5 | 8
  No | 11 | 10 | 7

10. Secondary Outcome: Opioid Dose Among Patients Receiving Opioids in the PACU
Description: Total opioid dose taken by patients who took any opioids in the PACU, measured in oral morphine equivalents (mg OME)
Time Frame: Duration of PACU stay (Average 2 hours)
Measure: Mean (Inter-Quartile Range); unit: mg OME
Arm/Group | FA Patients Under Popliteal Block + Spinal + Sedation | TSA Patients Under Brachial Plexus Block + General (LMA) | TSA Patients Under Brachial Plexus Block + Sedation
Number analyzed (Participants) | 4 | 5 | 8
mg OME | 22.5 [15 to 36.2] | 15 [10 to 19.5] | 18.9 [13.4 to 26.7]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during the period of enrollment and patient participation (Post-Operative Day 0 to Post-Operative Day 1).
Arm/Group | FA Patients Under Popliteal Block + Spinal + Sedation | TSA Patients Under Brachial Plexus Block + General (LMA) | TSA Patients Under Brachial Plexus Block + Sedation
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15

LIMITATIONS AND CAVEATS:
Limitations included generalizability, as the study was limited by anesthetic regimen, type of surgery, and patient population. We felt it was inappropriate to randomize general or spinal anesthesia for the purpose of this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes